CLINICAL TRIAL: NCT05241717
Title: Internet-Delivered Cognitive Behavioral Treatment for Chronic Pain in Adolescent Survivors of Childhood Cancer: A Single-group Feasibility Trial
Brief Title: WebMAP for Childhood Cancer Survivors
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Calgary (Other)
Responsible Party: Principal Investigator, Fiona Simone Maria Schulte, Associate Professor, University of Calgary
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HREBA.CC-21-0272
Record Dates: First submitted 2021-10-26; First posted 2022-02-16 (Actual); Last update posted 2022-05-18 (Actual); Status verified 2022-05

CONDITIONS: Chronic Pain; Survivorship; Childhood Cancer
MeSH Terms: conditions — Chronic Pain; Neoplasms

STUDY DESIGN:
Intervention Model Description: Mixed methods, single-arm feasibility study
Masking Description: All participants will be provided the intervention
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention arm (Experimental): All study participants will be given the intervention
  Interventions: Behavioral: Web-based Management of Adolescent Pain (WebMAP)

INTERVENTIONS:
Behavioral: Web-based Management of Adolescent Pain (WebMAP) — Participants will be asked to complete one module per week, which are approximately 20 minutes in length. Survivors and parents will be asked to spend approximately 4.5 hours each over the course of the intervention on WebMAP including 4 hours to complete the modules and 30 minutes total corresponding with a coach. Each week, patients log into WebMAP to learn a new skill and practice that skill for 1 week to allow time for skills acquisition. WebMAP consists of two separate, password-protected programs including one for adolescents and one for parents (http://webmap2.com).

SUMMARY:
Background: There are over 500,000 survivors of childhood cancer in North America alone. One in four survivors experiences chronic pain after treatment has completed. Youth with chronic pain report increased anxiety, depression, activity limitations, and sleep disturbances. An 8-week web-based cognitive-behavioral treatment for chronic pain (WebMAP) has demonstrated reduction in the pain in children but has not yet been explored in survivors. The objectives of the current study are to (1) test the feasibility and acceptability of WebMAP for a sample of survivors with chronic pain and their parents, (2) assess the acceptability of WebMAP using qualitative interviews, (3) assess WebMAP's effect on activity limitations, pain intensity, depression and anxiety symptoms, and sleep disturbances, and (4) assess WebMAP's effect on parent pain catastrophizing and parental response to their child's pain.

Methods: A single-arm mixed-methods pre-post intervention study design will be utilized. Participants will be 34 survivors and at least one of their parents/caregivers. Inclusion criteria are (1) cancer history (2) current age 11-17 years, (3) >2 years post-treatment or >5 years post-diagnosis, (4) pain present over prior 3 months impairing >1 area of daily life and occurring >1/month , (5) computer access with broadband internet. Survivors will complete a pre-treatment questionnaire, which will include: Child Activity Limitations Interview, the pain intensity Numerical Rating Scale, PROMIS - and Pain Interference, Anxiety, Depression, and Adolescent Sleep Wake Scale. Parents will complete the Pain Catastrophizing Scale - Parent Version and the Adult Responses to Child Symptoms. Upon completion of pre-treatment questionnaires (T0), survivors will begin WebMAP. After the 8 week intervention, survivors will complete the same measures (T1), and at 3 month follow-up (T2). Post-treatment interviews will be conducted to determine acceptability. Feasibility will be assessed via recruitment and retention rates. Treatment engagement will be measured by number of modules completed. Pre-post outcome data will be assessed using Linear Mixed Models. Qualitative data will be analyzed using thematic analysis. Patient and caregiver partners will be involved in study design, recruitment, interpretation of results, and knowledge translation.

Discussion: Investigating whether WebMAP is useful to survivors will be an important step in improving pain management in this population.

ELIGIBILITY:
Inclusion Criteria:

* history of any cancer diagnosis
* current age 11-17 years
* at least 2 years post-treatment or completed treatment and at least 5 years post-diagnosis
* pain present over prior 3 months that impairs at least one area of daily life and occurs at least 1/month
* computer access and literacy

Exclusion Criteria:

* not able to read/understand English
* developmental delays that would prevent them from completing the survey themselves or complete the intervention
* psychosis

Ages: 11 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 38 (Estimated)
Dates: Start 2022-06 (Estimated); Primary Completion 2023-07 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Feasibility assessed by the number of participants recruited | 1 year
  The number of participants recruited for the study will be part of the assessment of the feasibility of the trial.
Feasibility assessed by participant retention | 1 year
  The number of participants who complete the study will be part of the assessment of the feasibility of the trial.
Feasibility assessed by treatment adherence | 1 year
  The number of participants who complete at least 6 of the 8 modules of the intervention will be part of the assessment of the feasibility of the trial.
Acceptability of intervention assessed by a satisfaction survey | 3 months after the intervention
  A survey including open-ended questions will be created with patient partners to elicit feedback on specific modules. These questions will ask about what information was helpful and what may need to be adjusted to better serve youth with a history of cancer for both patients and parents. The satisfaction survey will be completed as part of the post-treatment questionnaire.
Feasibility, acceptability and satisfaction assessed by qualitative interviews | Immediately after the intervention
  Semi-structured interviews will be conducted with survivors upon treatment completion to assess feasibility, acceptability, and satisfaction with the program. Patient partners will be involved in creating the standard set of questions.
Satisfaction with intervention modules assessed by a satisfaction survey | 3 months after the intervention
  A survey including open-ended questions will be created with patient partners to elicit feedback on specific modules. These questions will ask about what information was helpful and what may need to be adjusted to better serve youth with a history of cancer for both patients and parents. The satisfaction survey will be completed as part of the post-treatment questionnaire.

SECONDARY OUTCOMES:
Pain intensity assessed by a pain rating | Baseline, immediatly after the intervention, 3 months after the intervention
  Daily surveys, administered through REDCap, will be used to assess daily presence of pain and pain intensity for 7 days at each assessment period. Pain intensity will be assessed with an item asking about the magnitude of pain experienced answered on an 11-point numerical rating scale (0 = no pain, 10 = worst pain). This measure of pain intensity has demonstrated to be a reliable and valid measure of pain in many populations of children 8 years and older (Baeyer et al., 2009; Castarlenas, Jensen, Baeyer, & Miro, 2017), but has not yet been validated in people with cancer.
Activity Limitations assessed by the Child Activity Limitations Interview | Baseline, immediatly after the intervention, 3 months after the intervention
  The Child Activity Limitations Interview is a measure of children's perceived difficulty in completing typical daily activities because of pain. The CALI will be collected for 1 week at each of the study timepoints. Survivors will choose the top 8 activities from a list of 21 and will be asked each day whether the activity occurred and how difficult the activity was to perform because of their pain. Difficulty ratings are measures on a five-point scale (0 = no difficulty, 4 = extremely difficult), with a range of zero to 32. Higher scores indicate greater functional limitations. Average daily limitation scores across each assessment period will be computed.
Anxiety and depressive symptoms and pain interference assessed by Patient Reported Outcomes Measurement Information System (PROMIS) measures | Baseline, immediatly after the intervention, 3 months after the intervention
  The PROMIS Anxiety and Depression instruments (Cook, Reeve, Ader, & Fries, 2010(31)) (8-item short form) will be administered via REDCap to screen for current symptoms of anxiety and depression. Survivors will complete the self-report instrument corresponding to their age (child: age 8-17; adult: age 18+). Items (e.g., "I felt worried") are rated on a five-point scale (1 = never, 5 = always). Higher scores signify greater severity of symptoms. Pain interference will be assessed using the four-item PROMIS interference scale for survivors 8-17 years of age, and the seven-item PROMIS interference scale for survivors over 18 years of age (Hinds et al., 2013). The PROMIS pediatric measures have been validated for use in pediatric oncology (Hinds et al., 2013).
Sleep quality assessed by the Adolescent Sleep Wake Scale | Baseline, immediatly after the intervention, 3 months after the intervention
  The Adolescent Sleep Wake Scale (ASWS-S) (32, 33) is a measure of the subjective perception of sleep quality. The ASWS-S is a 10-item measure where items representing symptoms of sleep disturbance are scored on a 6-point Likert scale (1 = always, 6 = never), and will be administered online via REDCap. The measure produces a total sum score where higher scores represent more severe sleep disturbance. The ASWS has demonstrated acceptable reliability and validity among populations of youth with comorbid sleep and medical conditions (34) and among ethnically diverse youth (33).
Catastrophizing about child's pain assessed by the Pain Catastrophizing Scale-Parent Version | Baseline, immediatly after the intervention, 3 months after the intervention
  The Pain Catastrophizing Scale - Parent Version (PCS-P) (37) is a 13-item measure used to assess parents' catastrophic thoughts and feelings about their child's pain and will be administered online via REDCap. Parents rate statements about their child's pain on a five-point Likert scale (i.e., "When my child has pain, I can't keep it out of my mind"). Items are summed to yield a total score and can also be summed to provide scores on three subscales: rumination, magnification, and helplessness. Lower scores indicate less catastrophizing. This scale has been found to have good reliability in parents with children who experience pain.
Parental responses to child's pain behaviors assessed by the Adult Responses to Children's Symptoms | Baseline, immediatly after the intervention, 3 months after the intervention
  The Adult Responses to Children's Symptoms (ARCS) (38, 39) measures parental responses to their child's pain behaviors and will be administered online via REDCap. The current study will only utilize the Protect subscale, which assesses parents' responses that either positively or negatively reinforce pain complaints. Parents' responses are rated on a five-point scale (0 = never, 4 = always). Subscale scores represent an average of the items, with higher scores indicating more frequent use of that behavioral style. This scale has demonstrated reliability and validity for use with parents of children with chronic pain (38, 39).
Parent distress assessed by the Kessler Psychological Distress Scale | Baseline, immediatly after the intervention, 3 months after the intervention
  The Kessler Psychological Distress Scale (40) is a 6-item measure used to assess non-specific psychological distress representing diagnoses of major depression and generalized anxiety disorder and also contains a positive affect domain. The measure has good precision in the 90-99th percentile range of the population, and has solid psychometric properties across major sociodemographic populations distribution in the United States of America and Canada (40). It also strongly discriminates between meeting and not meeting diagnostic thresholds for psychological disorders (40).

CONTACTS AND LOCATIONS:
Overall Officials: Fiona Schulte, PhD, Principal Investigator — University of Calgary
Locations (1):
- Alberta Children's Hospital, Calgary, Alberta, Canada

IPD SHARING:
Plan to Share IPD: Yes
All deidentified IPD will be provided upon request.
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: Data will be available after initial publication until 5 years after study completion.
Access Criteria: A .sps file of deidentified data will be shared upon request to the research contact.

REFERENCES:
- [Derived] Patton M, Carlson LE, Noel M, Palermo T, Forster V, Cho S, Schulte F. Internet-Delivered Cognitive Behavioral Treatment for Chronic Pain in Adolescent Survivors of Childhood Cancer: Protocol for a Single-Group Feasibility Trial. JMIR Res Protoc. 2023 Aug 1;12:e45804. doi: 10.2196/45804. PMID 37526959